CLINICAL TRIAL: NCT02332161
Title: Does Harvesting an Anterolateral Thigh (ALT) Flap Impact Lower Extremity Function and Activities of Daily Living (ADL) in Patients Undergoing Reconstructive Surgery for Head and Neck Cancer
Brief Title: Leg Function and ADL After ALT Reconstruction for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 13-1375
Record Dates: First submitted 2014-12-30; First posted 2015-01-06 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Free Tissue Flaps; Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: surveys, evaluative tests for leg function — See outcome measures

SUMMARY:
Anterolateral thigh (ALT) free flap tissue transfer is a commonly used method of head and neck reconstruction after head and neck cancer removal. The procedure involves removing some muscle, skin, and tissue from the thigh, and this may affect leg function. The purpose of this study is to determine the impact of ALT on ambulation and activities of daily living (ADLs)

DETAILED DESCRIPTION:
The ALT flap may be harvested as a subcutaneous, fasciocutaneous, musculocutaneous, or adipofascial flap. At our institution, three surgeons commonly use this method of free tissue transfer to reconstruct such defects. In our experience, patients following harvest of ALT flap have impairments in lower extremity function that result in decreased independence with transfers, gait and ability to independently perform ADLs. Consequently, these patients receive Physical and Occupational Therapy following surgery and a number of patients go on to receive therapy in a rehabilitation facility and/or as an outpatient. A number of studies have examined donor site morbidity and lower extremity function following ALT flap harvest. These studies, however, are heterogeneous and primarily use patient reported and non-standardized scales as outcome measures. Additionally, there is a paucity of literature related to Physical Therapy and Occupational Therapy outcomes and intervention with this patient population, despite frequent referral of these patients for post-surgical therapy.

This investigation will utilize the Lower Extremity Functional Scale, the Functional Independence Measure, dynamometry, video analysis of a single leg squat and walking speed in an effort to better assess the affect of ALT harvesting on patients' functional capacity post operatively. These tests are valid and reliable measures commonly utilized in Physical Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Over age 18;
2. Head and neck cancer;
3. To undergo anterolateral thigh free tissue transfer for head and neck reconstruction

Exclusion Criteria:

1. Inability to ambulate independently prior to surgery;
2. Inability to negotiate stairs prior to surgery;
3. Inability to follow simple commands;
4. Inability to negotiate stairs prior to surgery;
5. Previous free flap harvest from either lower extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient over age 18 undergoing anterolateral thigh free tissue transfer for head and neck cancer reconstruction at the University of Chicago
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Functional Scale | Pre- and Postoperative - subjects will be followed until discharge, and assessed again at 1 month follow-up
  The Lower Extremity Functional Scale (LEFS) is a validated self-report measure designed to assess the functional capabilities of patients with any lower extremity related musculoskeletal condition. Subjects will be assessed for a change from pre- to post-operative

SECONDARY OUTCOMES:
Lower Extremity Function | Pre- and Postoperative - subjects will be followed until discharge, and assessed again at 1 month follow-up
  Standing on one leg and walking, specifically duration of standing on one leg in minutes and distance walked up to 100 ft. Subjects will be assessed from pre-to-postoperative to determine the decline in leg function.
Functional Independence Measure | Pre- and Postoperative - subjects will be followed until discharge, and assessed again at 1 month follow-up
  The Functional Independence Measure (FIM) will assess subject ability to perform activities of daily living such as bathing, lower body dressing, toileting, bed to chair transfer, toilet transfer, walking on level and stairs, social interaction, problem solving and memory. We will assess the change from pre- to post-operative
Lower Extremity Strength | Pre- and Postoperative - subjects will be followed until discharge, and assessed again at 1 month follow-up
  Dynamometry will be performed in seated position to determine a change in muscle strength from pre- to post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Langerman, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543